CLINICAL TRIAL: NCT02094911
Title: Implementation and (Cost-)Effectiveness of Diabetes Prevention in Dutch Primary Health Care: From SLIM to SLIMMER
Brief Title: (Cost-)Effectiveness of SLIMMER Diabetes Prevention Intervention
Acronym: SLIMMER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wageningen University (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL37994.081.11
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Prevention; Combined lifestyle intervention; Primary health care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined lifestyle intervention (Experimental): Lifestyle counselling (nutrition and physical activity) by dietician and physiotherapist during 10-month intervention period
  Interventions: Behavioral: Combined lifestyle intervention
- Usual care group (Other): Subjects receive brochures on healthy lifestyle at baseline, and during the 10-month intervention period only usual care as provided by their own general practitioner.
  Interventions: Other: Usual care group

INTERVENTIONS:
Behavioral: Combined lifestyle intervention — 10-month intervention period with:
  * weekly group-based sports lessons supervised by a physiotherapist
  * individual dietary advice by a dietician
  * case management by practice nurse
  * maintenance programme to guide subjects to maintain lifestyle behaviour change
  Other Names: SLIMMER intervention
  Arms: Combined lifestyle intervention
Other: Usual care group — Written information on healthy lifestyle was provided at baseline, no individual advice or programme was provided. No additional appointments were scheduled, apart from the visits for follow-up measurements
  Arms: Usual care group

SUMMARY:
The overall aim of the project is to evaluate the (cost-)effectiveness of the SLIMMER diabetes prevention intervention in Dutch primary health care.

DETAILED DESCRIPTION:
This is a randomised controlled trial, conducted in a real-life setting (Dutch primary health care).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Impaired fasting glucose (IFG; i.e. venous plasma glucose concentration ≥6.1 and

  ≤6.9 mmol/l) during the past 5 years, according to the GP registration database OR diabetes risk score ≥7 as calculated from the Diabetes Risk Test
* Willing and able to participate in the intervention for at least 1.5 years
* Dutch speaking

Exclusion Criteria:

* Known diabetes mellitus
* Any chronic illness that makes 1.5-years survival improbable, interferes with glucose tolerance, or makes participation in a lifestyle intervention impossible
* Patients with any severe cardiovascular disease (this also includes history of cardiac dysrhythmia), unless GP gives agreement
* Medication known to interfere with glucose tolerance
* Any mental or physical disability that will hinder participation in the lifestyle intervention
* Severe psychiatric disease
* Patients who showed bad compliance in the past
* Participation in another regular vigorous exercise and/or diet programme, i.e.:

  * Intensive exercise programme: any exercise programme offered by a physiotherapist and/or patients sporting at least 3 times a week at their own initiative.
  * Intensive diet programme: patients who visited a dietician at least 3 times during the last year.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Change in fasting insulin | Baseline, end of intervention (12 months), after follow-up (18 months)

SECONDARY OUTCOMES:
Glucose tolerance | Baseline, end of intervention (12 months), after follow-up (18 months)
  fasting glucose, 2h glucose, 2h insulin, HbA1c
Serum lipids | Baseline, end of intervention (12 months), after follow-up (18 months)
  total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Body fatness | Baseline, end of intervention (12 months), after follow-up (18 months)
  body weight, BMI, waist and hip circumference, body fat
Physical fitness | Baseline, end of intervention (12 months), after follow-up (18 months)
  measured with six-minute walk test
Blood pressure | Baseline, end of intervention (12 months), after follow-up (18 months)
Medication use | Baseline, end of intervention (12 months), after follow-up (18 months)
Quality of Life | Baseline, end of intervention (12 months), after follow-up (18 months)
Eating behaviour | Baseline, end of intervention (12 months), after follow-up (18 months)
  Measured as nutrient intake and food intake, with a Food Frequency Questionnaire
Physical activity behaviour | Baseline, end of intervention (12 months), after follow-up (18 months)
  Measured with questionnaire
Behavioural determinants | Baseline, end of intervention (12 months), after follow-up (18 months)
  Determinants of nutrition and physical activity behaviour, measured with questionnaire
Process indicators | Baseline, end of intervention (12 months), after follow-up (18 months)
  Indicators to investigate how the intervention was delivered and received, measured with quantitative and qualitative methods

CONTACTS AND LOCATIONS:
Overall Officials: Edith Feskens, PhD, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] Duijzer G, Bukman AJ, Meints-Groenveld A, Haveman-Nies A, Jansen SC, Heinrich J, Hiddink GJ, Feskens EJM, de Wit GA. Cost-effectiveness of the SLIMMER diabetes prevention intervention in Dutch primary health care: economic evaluation from a randomised controlled trial. BMC Health Serv Res. 2019 Nov 11;19(1):824. doi: 10.1186/s12913-019-4529-8. PMID 31711499
- [Derived] den Braver NR, de Vet E, Duijzer G, Ter Beek J, Jansen SC, Hiddink GJ, Feskens EJM, Haveman-Nies A. Determinants of lifestyle behavior change to prevent type 2 diabetes in high-risk individuals. Int J Behav Nutr Phys Act. 2017 Jun 12;14(1):78. doi: 10.1186/s12966-017-0532-9. PMID 28606146
- [Derived] Duijzer G, Haveman-Nies A, Jansen SC, ter Beek J, Hiddink GJ, Feskens EJ. SLIMMER: a randomised controlled trial of diabetes prevention in Dutch primary health care: design and methods for process, effect, and economic evaluation. BMC Public Health. 2014 Jun 14;14:602. doi: 10.1186/1471-2458-14-602. PMID 24928217